CLINICAL TRIAL: NCT02252731
Title: A Phase 1, Open-label, One-sequence Crossover Study to Evaluate the Effect of Multiple Doses of FG 4592 on the Pharmacokinetics of Warfarin in Healthy Subjects
Brief Title: A Study to Evaluate the Effects of Multiple Doses of FG-4592 on the Exposure, Safety and Tolerability and Effect of Warfarin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1517-CL-0509; 2013-001043-31 (EudraCT Number)
Record Dates: First submitted 2014-06-10; First posted 2014-09-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Pharmacokinetics of FG-4592; Healthy Subjects
Keywords: Phase I; FG-4592; Warfarin; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — Warfarin; roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- warfarin and FG-4592 (Experimental): Single dose of warfarin and Multiple doses of FG-4592 in combination with a single dose of warfarin
  Interventions: Drug: Warfarin; Drug: FG-4592

INTERVENTIONS:
Drug: Warfarin — Oral
  Other Names: Coumadin®
Drug: FG-4592 — Oral
  Other Names: ASP1517,; roxadustat

SUMMARY:
This study will determine the effect of multiple doses of FG-4592 on the pharmacokinetics (PK) of a single dose of warfarin. It will evaluate the safety and tolerability of warfarin alone and in combination with multiple doses of FG-4592, and will evaluate the effect of multiple doses of FG-4592 on the pharmacodynamics (PD) of warfarin.

DETAILED DESCRIPTION:
The study consists of 2 periods, separated by a washout period (a minimum of 14 days after warfarin dosing on Day 1, Period 1). Screening takes place from Day -22 to Day -2.

Subjects are admitted to the clinical unit on Day -1 of Period 1. On Day 1 of the first period, subjects receive a single oral dose of warfarin. After completion of all assessments on Day 8, subjects are discharged from the clinical unit on the condition that there are no medical reasons for a prolonged stay. They return to the clinical unit on Day -1 of the second period, after the washout period.

In Period 2, the subjects receive multiple doses of FG 4592. On Day 7 of Period 2, FG 4592 is given concomitantly with warfarin. After completion of all assessments on Day 16 of Period 2, subjects are discharged from the clinic on the condition that there are no medical reasons for a prolonged stay. The subjects return for an End of Study Visit (ESV) 5 to 9 days after the last assessment of Period 2 (or after early withdrawal).

Safety assessments are performed throughout the study. Blood and urine samples are collected for PK and PD assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male subject and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of two forms of birth control.
* Male subject must not donate sperm starting at screening and throughout the study period and for 90 days after the final study drug administration.
* Female subject must be either of non-childbearing potential or, if of childbearing potential, must have a negative pregnancy test at screening and Day -1 and must use two forms of birth control.
* Female subject must not donate ova starting at screening and throughout the study period and for 28 days after the final study drug administration.

Exclusion Criteria:

* Subject has a known or suspected hypersensitivity to FG 4592, warfarin, or any components of the formulations used.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to admission to the clinical unit [Day -1].
* Subject is lactose intolerant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
PK of S-warfarin and R-warfarin in plasma measured by area under the curve from the time of dosing extrapolated to time infinity (AUCinf) | Period 1 (Day 1 to Day 8); Period 2 (Day 7 to Day 16)
PK of S-warfarin and R-warfarin in plasma measured by maximum concentration (Cmax) | Period 1 (Day 1 to Day 8); Period 2 (Day 7 to Day 16)

SECONDARY OUTCOMES:
PK profile of S-warfarin and R-warfarin in plasma | Period 1 (Day 1 to Day 8); Period 2 (Day 7 to Day 16)
  area under the concentration-time curve from the time of dosing to the last measurable concentration (Clast) (AUClast), unbound AUC from the time of dosing to Clast (AUClast,u), AUC from the time of dosing extrapolated to time infinity (AUCinf), unbound AUC extrapolated to infinity (AUCinf,u), maximum unbound plasma concentration (Cmax,u), apparent total body clearance after extra-vascular dosing (CL/F), unbound apparent total body clearance after extravascular dosing (CLu/F), fraction unbound (fu), time interval between the time of dosing and the first measurable concentration (tlag), time of the maximum concentration (tmax), terminal elimination half-life (t1/2), apparent volume of distribution during the terminal elimination phase after single extravascular dosing (Vz/F), unbound apparent volume of distribution during terminal phase after oral administration (Vz,u/F)
PK profile of FG-4592 in plasma | Period 2 (Day 1 to Day 15)
  AUC from time point 0 to time point 24 hours (AUC0-24h), AUClast, AUCinf , Cmax, concentration at pre-dose for repeated dosing (Ctrough), tmax, t1/2, CL/F, and Vz/F
PK profile of FG-4592 in urine | Period 2 (Day 7 to Day 8)
  renal clearance (CLR), unbound CLR from time point 0 to 24 hours (CLR,0-24h), cumulative amount of drug excreted unchanged into urine from time of dosing extrapolated to time infinity (Aeinf), percent of drug excreted unchanged into urine from time of dosing extrapolated to time infinity in percent of dose (Aeinf%), cumulative amount of drug excreted unchanged into urine, from time of dosing up to the collection time of the last measurable concentration (Aelast), percent of drug excreted into urine from time of dosing up to the collection time of the last measurable concentration in percent of dose (Aelast%), cumulative amount of drug excreted unchanged into urine, from time of dosing up to the collection time of 24 hours (Ae0 24h), cumulative amount of drug excreted unchanged into urine, from time of dosing up to the collection time of 24 hours in percent of dose (Ae0-24h%)
Pharmacodynamics profile of warfarin in plasma | Period 1 Day 1 to to ESV (5 to 9 days after the last protocol defined assessment of Period 2 (or after early withdrawal))
  area under the Prothrombin Time (PT)-time curve from the time of dosing until the last sample collected (AUCPT,last), maximal PT (PTmax), time to reach PTmax (tPT,max), area under the International Normalized Ratio (INR)-time curve from the time of dosing until the last sample collected (AUCINR,last), maximal INR after Drug Administration (INRmax), time to reach the INRmax (tINR,max)
Safety profile | Screening (Day -22 to Day -2) to ESV (5 to 9 days after the last protocol defined assessment of Period 2 (or after early withdrawal))
  Safety profile includes Adverse Events (AEs), vital signs, physical examination, laboratory tests, electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Parexel International GmbH, Berlin, Germany

REFERENCES:
- [Derived] Groenendaal-van de Meent D, den Adel M, Rijnders S, Krebs-Brown A, Kerbusch V, Golor G, Schaddelee M. The Hypoxia-inducible Factor Prolyl-Hydroxylase Inhibitor Roxadustat (FG-4592) and Warfarin in Healthy Volunteers: A Pharmacokinetic and Pharmacodynamic Drug-Drug Interaction Study. Clin Ther. 2016 Apr;38(4):918-28. doi: 10.1016/j.clinthera.2016.02.010. Epub 2016 Mar 4. PMID 26947173